CLINICAL TRIAL: NCT03097536
Title: Migraine and Homeostasis:What Can we Learn From Glucose
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 impact
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Alexandra Hovaguimian, Instructor in Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000419
Record Dates: First submitted 2016-07-12; First posted 2017-03-31 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Migraine Headache
Keywords: Blood Sugar
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luna Bar Intervention (Experimental): Participants will be asked to monitor their blood sugar during migraine. Study data will also include blood glucose levels, pain severity, 24-hour food diary, 24-hour exercise diary, duration of sleep, perception of quality of sleep, and last menstrual period. This information will be recorded at times when a Luna bar is not consumed, and at times when a Luna Bar is consumed. Participants will serve as their own controls.
  Interventions: Other: Luna Bar
- Morning Migraine (No Intervention): Participants will be asked to monitor their blood sugar on headache free days as well as during migraine. This arm is only for participants who identify as having morning migraine. Study data will also include blood glucose levels, pain severity, 24-hour food diary, 24-hour exercise diary, duration of sleep, perception of quality of sleep, and last menstrual period. Participants will serve as their own controls.

INTERVENTIONS:
Other: Luna Bar — Luna Bar (blueberry bliss or lemon zest flavor) product of Clif
  Arms: Luna Bar Intervention

SUMMARY:
Patients with migraine often report that stressors such as skipping a meal can bring on a migraine whereas some patients report that their migraine improves with food. Few studies to date have looked at the relationship between blood glucose (sugar) and migraine. We are conducting this study to better understand whether or not changes in blood glucose levels can trigger migraine or provide relief during a migraine attack.

DETAILED DESCRIPTION:
The purpose of this pilot and feasibility study is to assess if changes in blood glucose both trigger migraine and can provide analgesia. This information will provide a vital basis for the mechanism of migraine and offer insights into better treatments as well as prevention.

This is a pilot unblinded randomized trial with two independent components, Aims 1 and 2. It is not possible to blind the current protocol both in terms of the blood sugar readings and the luna bar, non-luna bar intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, age 18-65 with episodic migraine with or without aura (ICHD-II) and/or morning onset and/or patients who self identify that eating reduces their migraine intensity.

Exclusion Criteria:

* Chronic migraine, use of hypoglycemic medication, DM I or II, abnormal finger stick glucose, obesity, comorbid eating disorders, pregnancy, seizure disorder, other serious mental or physical condition that would impair participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
The difference in blood glucose on days with migraine compared to blood glucose on days without migraine | Change Measure: migraine days and non-migraine days over 3 month period.
  The primary endpoint will be the difference in blood glucose on days with migraine compared to blood glucose on days without migraine using repeated measure ANOVA

SECONDARY OUTCOMES:
The primary outcome is the change in pain score from the time of pain plateau to the pain score at 120 minutes as measured by a visual analogue scale. | Change Measure: migraine days and non-migraine days over 3 month period.
  The primary outcome is the change in pain score from the time the patients pain plateaus (as measured by having a stable pain score for 60 minutes) compared to the pain score at 120 minutes using a repeated measures ANOVA. We will compare these measures on migraine days with Luna and without Luna bar (control days) using a repeated measures ANOVA

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Hovaguimian, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medial Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided